CLINICAL TRIAL: NCT03324399
Title: A Study of Protein Metabolism, Microbiome and Investigational Probiotic Use in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Study of Protein Metabolism, Microbiome and Investigational Probiotic Use in Patients With ALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIHG-2017.004-ALS
Record Dates: First submitted 2017-09-05; First posted 2017-10-27 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
Keywords: ALS; Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Amino Acid levels (Experimental): Comparison between high amino acid levels and low amino acid levels of clinical global assessments, muscle strength and spasticity and functional assessments.
  Patients taking proprietary probiotic
  Interventions: Dietary Supplement: probiotic
- Low Amino Acid levels (Experimental): Comparison between high amino acid levels and low amino acid levels of clinical global assessments, muscle strength and spasticity and functional assessments.
  Patients taking proprietary probiotic
  Interventions: Dietary Supplement: probiotic

INTERVENTIONS:
Dietary Supplement: probiotic — a proprietary probiotic formulation

SUMMARY:
ALS, also known as "Lou Gehrig's" disease, is a neurodegenerative disease which is fatal. Treatment for ALS is limited and currently consists of primary symptom relief or support. In addition, time from diagnosis to death averages 3-5 years. New Biotic, LLC has submitted an Orphan Drug Designation Application for an investigational probiotic and have indicated the need for more study of this orphaned drug in ALS patients.

DETAILED DESCRIPTION:
This will be an exploratory protocol of 10 patients and expect to screen approximately 25-30 patients.

The purpose of our study is to examine amino acid levels in plasma pre and post prandial as well as longitudinal gut microbiome in ALS patients taking the investigational probiotic.

1. Purpose: Evaluate the clinical outcomes of muscle strength, clinical global assessments and spasticity in patients taking an Investigational probiotic.
2. Measure changes in questionnaires relating to subjective functional assessments, quality of life, and pain levels over 24 weeks.
3. Describe plasma amino acid levels before and after a protein food challenge in ALS patients of spinal and bulbar type.
4. Evaluate and describe the gut microbiome of patients with ALS.

Design:

This is a non-randomized, open-label, two-group pilot study of plasma amino acid levels, gut microbiome, and of investigational probiotic use in patients with ALS. Participants will be placed into two groups based on certain post-prandial amino acid levels. Patients will be stratified for eligibility based on the results of their amino acid profiles.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sporadic ALS, definite or probable disease,-revised El Escorial criteria
* Patient must be able to understand the purpose and procedures of the study, sign informed consent and comply with requirements of the protocol.
* Age 18 and older.
* Normal serum Magnesium (1.7 - 2.3 mg/dL) and Manganese (4.7 - 18.3 ng/mL) levels or adequate supplement to obtain normal serum Mg (if Manganese levels are low (<1.7 mg/dL), Hair Manganese will be evaluated before starting probiotic, and inclusion to the protocol will be at the principal investigators discretion).

Exclusion Criteria:

* Need for consumption of frequent antibiotics, gut pH increasing medications, and/or alkaline water.
* Patient unable to maintain regular follow up or submit to informed consent
* Stool pH >7.5 - The ideal stool pH for growth and function of the investigational probiotic is 6-6.5.
* Patients who are judged to be ineligible for study entry by investigator or sub-investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Evaluate amino acid levels before and after probiotic use. | 6 months
  Amino acid profiles will be compared before the probiotic use and over a period of treatment for 6 months.

SECONDARY OUTCOMES:
Measure changes in questionnaires relating to subjective functional assessments. | 6 months
  Changes will be measured with Amyotrophic Lateral Sclerosis -Functional Rating Scale (ALS-FRS).
  The ALS-FRS is a 12 item questionnaire to assess bulbar, limb, and respiratory functions. The scores may range from 0, which is the worst function, to 48 which is the best function. This questionnaire is self-administered, and can be completed with assistance from a family member. The scores range from 0-48. The highest scores reflect no changes, or difficulty with tasks assessed. Low scores indicate poor functioning and need for assistance.
Measure changes in Quality of Life. | 6 months
  Changes will be measured with the Amyotrophic Lateral Sclerosis -Quality of Life questionnaire. The ALS-QOL is a 50-item, self-administered, questionnaire which includes 7 scores. These scores represent six domains and a total average score. The six domains are 1) Negative Emotion, 2) Interaction, 3) Intimacy, 4) Religiosity, 5) Physical and 6) Bulbar.
Evaluate pain levels with the Numbered Pain Scale. | 6 months
  Changes in pain rating of 0 - 10 will be collected during the 6 months of study.

CONTACTS AND LOCATIONS:
Overall Officials: Francine Arneson, MD, Principal Investigator — Avera Medical Group Palliative Medicine Sioux Falls
Locations (1):
- Avera Medical Group Palliative Medicine Sioux Falls, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No